CLINICAL TRIAL: NCT05764057
Title: DAPAgliflozine to Attenuate Cardiac RemOdeling afTEr aCuTe myOcardial Infarction
Acronym: DAPAPROTECTOR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP211054; 2022-001901-28 (EudraCT Number); AOM20806 (Other Grant/Funding Number: Other Grant/Funding Number)
Record Dates: First submitted 2023-03-01; First posted 2023-03-10 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: AMI; STEMI; NSTEMI; Left Ventricular Dysfunction
Keywords: Acute myocardial infarction; Left ventricular dysfunction; Dapagliflozin; Transthoracic echocardiography; Cardiac remodeling; Cardiovascular Intensive Care Unit (CICU)
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Ventricular Dysfunction, Left | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin 10mg daily + standard of care (Experimental): Dapagliflozin 10mg per day will be administered orally, as in clinical practice
  Interventions: Drug: Dapagliflozin propanediol (FORXIGA™/FARXIGA™1)
- Placebo + standard of care (Placebo Comparator): Placebo will be administered orally
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Dapagliflozin propanediol (FORXIGA™/FARXIGA™1) — Dapagliflozin (10 mg per day; per os) on top of standard of care as recommended in current guidelines* for 6 months (experimental group)
  *All patients will receive optimal medical therapy (including antithrombotic, beta-blockers, statins, angiotensin converting enzyme inhibitors or angiotensin receptor blocker or sacubitril/valsartan, diuretics, antagonists of the mineralocorticoid receptor) according to their clinical condition as recommended.
  Arms: Dapagliflozin 10mg daily + standard of care
Drug: Placebo comparator — Placebo daily on top of standard of care as recommended in current guidelines* for 6 months (control group)
  *All patients will receive optimal medical therapy (including antithrombotic, beta-blockers, statins, angiotensin converting enzyme inhibitors or angiotensin receptor blocker or sacubitril/valsartan, diuretics, antagonists of the mineralocorticoid receptor) according to their clinical condition as recommended.
  Arms: Placebo + standard of care

SUMMARY:
Recent clinical trials have proven the cardiovascular benefits of new medications for patients with heart failure with reduced ejection fraction (HFrEF), especially sodium-glucose co-transporter 2 (SGLT2) inhibitors. There are no existing randomized clinical trials evaluating the efficacy and safety of dapagliflozin (nor any other SGLT2-inhibitor) to limit cardiac remodeling in patients with acute myocardial infarction (AMI) and left ventricular (LV) dysfunction.

Preventing cardiac remodeling, an established predictor of subsequent heart failure (HF) and cardiovascular death, is likely to translate into benefit in reducing clinical events in post-MI patients.

DETAILED DESCRIPTION:
DAPA-PROTECTOR is a prospective multicenter, randomized, double blind, phase III trial.

Patients with confirmed AMI (e.g., STEMI or very high-risk NSTEMI) with LV dysfunction (LVEF≤45%) after completion of percutaneous coronary intervention (PCI) will be assessed for eligibility. Patients will be randomized (in a 1:1 ratio) to receive dapagliflozin (10mg once day) or placebo for 6 months, on top of standard of care as recommended in current guidelines. Treatment will be prescribed as soon as possible after admission The first TTE (TTE-1) will be performed to confirm inclusion criteria (LVEF≤45%). Four visits are scheduled: at baseline and randomization (Visit D0), at discharge from the CICU (Visit 2) at Month 3 ±2 weeks (Visit 3), and at Month 6 (+ 4 weeks) (Visit 4). After randomization, Visit 2 and Visit 3 will be scheduled to check the tolerance of the drug. In addition, a phone call will be done to the patient to make sure he's not taking any Dapagliflozin (or equivalent as Empagliflozin) in addition to experimental treatment. Finally, the last visit (Visit 4) will be scheduled to collect clinical follow-up and to perform a TTE (TTE-2). Efficacy criteria will be assessed from randomization to Month 6 by TTE. All TTE results will be anonymized and centralized at a Corelab with assessment by independent cardiologists unaware of the patient treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* STEMI (e.g., ST elevation above the J-point of ≥0.1 millivolt in ≥two contiguous leads or left bundle branch block) or very high-risk NSTEMI (e.g., dynamic ECG changes or ongoing chest pain or acute heart failure or hemodynamic instability independent of ECG changes or life-threatening ventricular arrhythmias) with LV dysfunction (LVEF ≤45%); after completion of PCI or angiography procedure
* eGFR ≥ 25 mL/Min per 1.73m²;
* Systolic blood pressure (SBP) before first dosing >100 mmHg and/or Diastolic blood pressure (DBP) >70 mmHg before first dosing;
* Ability to provide written informed consent and willing to participate in the 6-month follow-up period.
* Affiliation to a national health care system (AME are not allowed).

Exclusion Criteria:

* Cardiogenic shock (SBP <90 mmHg with clinical signs of low output or patients requiring inotropic agents) at randomization;
* Referred to surgery for coronary artery bypass grafting (CABG) or treatment of acute complications (e.g. ventricular septal rupture);
* Any other form of diabetes than diabetes type 2
* History of diabetic ketoacidosis (DKA); Known contra-indication to SGLT-2 inhibitors (hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption);
* >1 episode of severe hypoglycemia within the last 6 months under treatment with insulin or sulfonylurea;
* Acute symptomatic urinary tract infection (UTI) or genital infection at the time of randomization;
* Concomitant treatment (and/or within the 4 weeks prior to the baseline visit) with any SGLT-2 inhibitor (dapagliflozin, canagliflozin, empagliflozin)
* Echocardiographic examination of insufficient quality to permit adequate analysis of the study end-points.
* Impossibility to evaluate cardiac remodeling using TTE (e.g., pacemaker or defibrillator …);
* Atrial fibrillation rhythm at randomization;
* Life expectancy <6 month;
* Known pregnancy at time of randomization;
* Breastfeeding women
* Females of childbearing potential without adequate contraceptive methods (i.e. sterilization, intrauterine device, vasectomized partner; or medical history of hysterectomy)
* Current participation in another interventional trial. Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-10-12 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction (LVEF) from baseline to Month 6 (±1 month) by TTE | 6 months (+4 weeks) from randomization
  Two primary endpoints will allow to evaluate two independent and potent predictors of mortality after AMI: 1) Cardiac systolic function, assessed by change in left ventricular ejection fraction (LVEF) from baseline to Month 6 (+4 weeks) ) by TTE; 2) Remodeling, assessed by change in left atrium volume (LAV) from baseline to Month 6 (+4 weeks) by TTE.
Change in left atrium volume (LAV) from baseline to Month 6 (±1 month) by TTE | 6 months (+4 weeks) from randomization
  Two primary endpoints will allow to evaluate two independent and potent predictors of mortality after AMI: 1) Cardiac systolic function, assessed by change in left ventricular ejection fraction (LVEF) from baseline to Month 6 (+4 weeks) ) by TTE; 2) Remodeling, assessed by change in left atrium volume (LAV) from baseline to Month 6 (+4 weeks) by TTE.

SECONDARY OUTCOMES:
Change in left ventricular end-systolic volume (LVESV) | 6 months (+4 weeks) from randomization
  Comparison in each group from baseline to Month 6 (±1 month) using TTE. To assess the efficacy and safety of dapagliflozin compared to placebo in addition to optimal secondary prevention in the prevention of cardiac dysfunction after AMI with LV dysfunction.
Change in left ventricular end-diastolic volume (LVEDV) | 6 months (+4 weeks) from randomization
  Comparison in each group from baseline to Month 6 (+4 weeks) using TTE. To assess the efficacy and safety of dapagliflozin compared to placebo in addition to optimal secondary prevention in the prevention of cardiac dysfunction after AMI with LV dysfunction.
Change in LV global longitudinal strain (LS) | 6 months (+4 weeks) from randomization
  Comparison in each group from baseline to Month 6 (+4 weeks) using TTE. To assess the efficacy and safety of dapagliflozin compared to placebo in addition to optimal secondary prevention in the prevention of cardiac dysfunction after AMI with LV dysfunction.
Change in left atrial strain (LAS) | 6 months (+4 weeks) from randomization
  Comparison in each group from baseline to Month 6 (+4 weeks) using TTE. To assess the efficacy and safety of dapagliflozin compared to placebo in addition to optimal secondary prevention in the prevention of cardiac dysfunction after AMI with LV dysfunction.
Duration of hospital stay (index hospitalization) | 6 months (+4 weeks) from randomization
  Comparison between both groups (experimental vs. placebo) To assess the efficacy and safety of dapagliflozin compared to placebo in addition to optimal secondary prevention in the prevention of cardiac dysfunction after AMI with LV dysfunction.
All-cause mortality at 6-months | 6 months (+4 weeks) from randomization
  Comparison between both groups (experimental vs. placebo) Comparison between both groups (experimental vs. placebo) To assess the efficacy and safety of dapagliflozin compared to placebo in addition to optimal secondary prevention in the prevention of cardiac dysfunction after AMI with LV dysfunction
Cardiovascular death or worsening HF at 6-months | 6 months (+4 weeks) from randomization
  Comparison between both groups (experimental vs. placebo) To assess the efficacy and safety of dapagliflozin compared to placebo in addition to optimal secondary prevention in the prevention of cardiac dysfunction after AMI with LV dysfunction
Number of re-admission due to HF at 6-months | 6 months (±1 month) from randomization
  Comparison between both groups (experimental vs. placebo) To assess the efficacy and safety of dapagliflozin compared to placebo in addition to optimal secondary prevention in the prevention of cardiac dysfunction after AMI with LV dysfunction
Change from baseline to Month 6 (+4 weeks) in LVESV, LVEDV, LAV, LVEF, LV global LS, LAS and pulmonary congestion (normal lung, mild, moderate or severe ultrasound lung comets [ULCs]) using TTE at month 6 | 6 months (+4 weeks) from randomization
  Comparison between both groups (experimental vs. placebo) To assess the efficacy and safety of dapagliflozin compared to placebo in addition to optimal secondary prevention in the prevention of cardiac dysfunction after AMI with LV dysfunction
Change from baseline to Month 6 (+4 weeks) in plasma levels of NT-pro BNP and HBA1C | 6 months (+4 weeks) from randomization
  Comparison between both groups (experimental vs. placebo) To assess the efficacy and safety of dapagliflozin compared to placebo in addition to optimal secondary prevention in the prevention of cardiac dysfunction after AMI with LV dysfunction
Change in body weight from baseline to Month 6 (+4 weeks) | 6 months (+4 weeks) from randomization
  Comparison between both groups (experimental vs. placebo) To assess the efficacy and safety of dapagliflozin compared to placebo in addition to optimal secondary prevention in the prevention of cardiac dysfunction after AMI with LV dysfunction
Adverse events | 6 months (+4 weeks) from randomization
  Comparison between both groups (experimental vs. placebo) of Adverse events with particular focus to those potentially related to dapagliflozin complications (e.g., all symptoms of volume depletion, major hypoglycemia, genital infections, diabetes ketoacidosis, changes in liver function parameters [ASAT, ALAT ≥3 USN].
  To assess the efficacy and safety of dapagliflozin compared to placebo in addition to optimal secondary prevention in the prevention of cardiac dysfunction after AMI with LV dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne PUYMIRAT, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Cardiology AP-HP Hôpital européen Georges - Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided